# A Development Study to Evaluate a Nasal Mask for the Treatment of Obstructive Sleep Apnea

NCT04011826

**DATE: 17 October 2019** 



# **Clinical Investigation Plan**





This page intentionally left blank

### Table of Contents

| 1. | Revision | on History | 5 |
|---|---|---|---|
| | 1.1. | List of Abbreviations | 5 |
| 2. | Docum | ent Information | 6 |
| | 2.1. | Purpose and Scope | 6 |
| | 2.2. | Confidentiality Statement | 6 |
| | 2.3. | Persons Authorized to Amend the CIP | . |
| | 2.4. | Monitoring Arrangements | 6 |
| | 2.5. | Data Management | 7 |
| 3. | Investi | gator Information | 7 |
| | 3.1. | Principal Investigator | 7 |
| | 3.2. | Coordinating Investigator | 7 |
| | 3.3. | Other Investigators | . |
| | 3.4. | Institution | 8 |
| 4. | Sponso | or Information | 8 |
| | 4.1. | Primary Sponsor Details | 8 |
| | 4.2. | Overseas Representative | . |
| 5. | Device | Information | 9 |
| | 5.1. | Identification of the Medical Device | g |
| | 5.2. | Device Risk Analysis and Management | g |
| 6. | Justific | cation for a Clinical Trial | 10 |
| | 6.1. | Synopsis | 10 |
| | 6.2. | Literature Review | 11 |
| | 6.3. | Preclinical Testing | 11 |
| | 6.4. | Previous Clinical Experience | 11 |
| | 6.5. | Justification for Administration | 12 |
| 7. | Objecti | ves of the Clinical Investigation | 12 |
| | 7.1. | Hypothesis | 12 |
| | 7.2. | Objectives | 12 |
| | 7.3. | Population | 12 |
| | 7.4. | Risks | 13 |
| | 7.5. | Essential Requirements of the Relevant Directive | 13 |
| 8. | Clinica | I Investigation Design | . |
| | 8.1. | Type of Investigation | 13 |
| | 8.2. | Controls | 14 |
| | 8.3. | Bias | 14 |
| | | End Points | |
| | | 4.1. Primary Outcome | |
| | 8. | 4.2. Secondary Outcomes | 14 |

| | 8.5. Variables | 14 |
|---|---|---|
| | 8.6. Measurements | |
| | 8.7. Equipment | 17 |
| | 8.8. Inclusion / Exclusion criteria | |
| | 8.9. Point of Enrolment | 18 |
| | 8.10. Patient Procedure | 18 |
| | 8.11. Withdrawal Criteria | 25 |
| | 8.12. Number of Trial Subjects | 25 |
| | 8.13. Follow up Plan | 25 |
| | 8.14. Foreseeable Complications | 26 |
| 9. | Clinical Trial Documentation | |
| | 9.1. Consent and Recruitment | |
| | 9.2. Case Report Form | |
| | 9.2.1. Case Report Form Signatories | |
| | 9.3. Insurance Statement | |
| | 9.4. Record of Deviations | |
| STA: | TISTICAL CONSIDERATIONS | 26 |
| O I A | 9.5. Description of the Statistical Design | |
| | 9.6. Sample Size | |
| | 9.7. Pass/Fail Criteria | |
| | 9.8. Statistical Termination | |
| | 9.9. Statistical Procedure Deviations | |
| | 9.10. Selection Criteria | 28 |
| | 9.11. Statistical Data Management | 28 |
| 10. | Adverse Events and Termination | |
| 10. | 10.1. Emergency Contact Details | |
| | 10.2. Foreseeable Adverse Events | |
| | 10.3. Reporting Adverse Events | |
| | 10.4. Early Termination | |
| | 10.4.1. Investigator | |
| | 10.4.2. Sponsor | 30 |
| | 10.4.3. Institutional Review Board (IRB) or Independent E | |
| | · , , · · | , , |
| 11. | Publication Policy | 30 |
| 12. | Approval | 30 |
| 13. | References | 32 |
| 14. | Appendix A: Recruitment Script | |
| | Detailed Information for each Visit (if requested) | |
| 15. | Appendix B: Participant Questionnaire | |
| 16. | | |

17. Appendix D: Researcher Questionnaire......

# 1. Revision History

| Revision | Date |
|----------|--------------------|
| Α | 11 June 2019 |
| В | 10 July 2019 |
| C | 17 October<br>2019 |

### 1.1. List of Abbreviations

AE Adverse Event

AHI Apnea Hypopnea Index

APAP Automatic Positive Airway Pressure

BPAP Bi-Level Positive Airway Pressure

CIA Clinical Investigation Administration

CIP Clinical Investigation Plan

CPAP Continuous Positive Airway Pressure

CRF Case Report Form

CSI Clayton Sleep Institute

F&P Fisher & Paykel Healthcare

GCP Good Clinical Practice

HA Hazard Analysis

IB Investigators Brochure

ICF Informed Consent Form

ICH International Conference on Harmonization of Technical Requirements for

Registration of Pharmaceuticals for Human Use

IRB Independent Review Board

| OSA | Obstructive Sleep Apnea |
|-----|--------------------------|
| PAP | Positive Airway Pressure |
| SAE | Serious Adverse Event |
| SME | Subject Matter Expert |
| UI | User Instructions |

### 2. **Document Information**

### 2.1. **Purpose and Scope**

The purpose of the trial is to evaluate the performance, comfort and ease of use (usability) of the F&P Nasal mask in the home environment in regards to satisfaction.

### 2.2. **Confidentiality Statement**

This document contains confidential information belonging to Fisher & Paykel Healthcare and is provided for the sole purpose of enabling an evaluation of a possible collaboration with Fisher & Paykel Healthcare to undertake the proposed clinical research. This document must be maintained in a confidential manner at all times and any disclosure, distribution or reproduction of this document outside the intended purpose is prohibited.



### 2.4. **Monitoring Arrangements**

F&P will be conducting the study, and as such the investigators will monitor the progress of the investigation. Planned monitoring activities will take place at Visit 1, 2 and 3 by a F&P Clinical Researcher as well as once during the course of the study extension as outlined below:





The principal investigator will have access to all source documents needed to verify the entries on the Case Report Forms (CRF) and other protocol- related documents; provided that participant confidentiality is maintained in agreement with local regulations. It will be the principal investigator's responsibility to inspect the CRF at regular intervals throughout the investigation, to verify the adherence to the protocol and the completeness, consistency and accuracy of the data being entered on them.

The investigator's file will contain the protocol/amendments, financial disclosure form, CRFs, data clarification and query forms, Independent Review Board (IRB) approval with correspondence, informed consent, staff curriculum vitae and authorization forms, screening and enrolment logs, and other appropriate documents/correspondence as per International Conference on Harmonization (ICH) and Good Clinical Practice (GCP) and local regulations.

### 2.5. Data Management

Data obtained for this investigation will be recorded in source documents and attached to the CRF for both the administration of the study and collection of participant data.

Original CRFs will be stored for 15 years by Fisher & Paykel Healthcare. Original Informed Consent Forms and copies of the CRF will be stored on site at Clayton Sleep Institute (CSI) for 15 years.

## 3. Investigator Information

### 3.1. Principal Investigator

Name: Mark Muehlbach

Address: 2531 S Big Bend Blvd, Maplewood, MO 63143, USA

Phone: 314-645-5855

Professional Position: Clinical Director

### 3.2. Coordinating Investigator

Name: Mr. Matthew Lee Uhles

Address: 2531 S Big Bend Blvd, Maplewood, MO 63143, USA

Email: uhlesm@claytonsleep.com

Phone: 314-645-5855 Ext 318

Professional Position: Chief Operating Officer



### 3.4. Institution

Name: Clayton Sleep Institute

Address: 2531 S Big Bend Blvd, Maplewood, MO 63143, USA

Email: uhlesm@claytonsleep.com

Phone: 314-645-5855

Country of residence: United States of America

# 4. Sponsor Information

### 4.1. Primary Sponsor Details

Name of Business: Fisher & Paykel Healthcare Limited

Address: 15 Maurice Paykel Place, East Tamaki, Auckland, New Zealand.

Name of Sponsor contact person: Bhavi Ogra

Phone: +64 9 574 0123 Ext 7882 Email: <a href="mailto:bhavi.ogra@fphcare.co.nz">bhavi.ogra@fphcare.co.nz</a>

Profession: Clinical Research Manager

Country of residence: New Zealand



### 6. Justification for a Clinical Trial

### 6.1. Synopsis

The investigation is a prospective, non-randomized, non-blinded study. This investigation is designed to evaluate the performance (leak and comfort) as well as participant's overall acceptance of the F&P Nasal mask amongst participants with diagnosed OSA. A minimum of 45 participants with OSA currently using a nasal, sub-nasal and/or pillows mask will be recruited by CSI. The phone recruitment script is available in Appendix A. CSI will recruit all participants within three weeks of beginning of the study.

This study will involve a baseline visit (Visit 1) where participants' informed consent for the F&P Nasal mask trial (CIA-262) will be gained. The participant's prescribed PAP therapy treatment settings will be gathered as well. Participants will also fill out a questionnaire (Appendix B) to gain a better understanding of their satisfaction of their current mask.

Visit 2 will take place  $7 \pm 3$  days after Visit 1. At this visit, participants will be fitted with the F&P Nasal mask and will be asked a few questions in the form of a structured questionnaire. Initial impressions, comments and photographs will be captured via recorded audio and video (provided the participant has given consent). If the participant does not provide video and/or audio consent, only written notes will be taken. Baseline efficacy data will be downloaded from participants' PAP/BPAP therapy devices. Participants will also be issued a sleep diary (Appendix C) to record daily feedback of the Nasal mask.

A follow up phone call will be made by CSI 3±1 days after Visit 2 and feedback will be recorded in the CRF.

Visit 3 will take place  $14 \pm 3$  days after Visit 2. The participants will return to the site and provide their feedback on the F&P Nasal mask in the form of verbal comments and a structured questionnaire (Appendix B and D). Photographs will be captured as well as audio and video will be recorded during this visit (provided the participant has given consent). If the participant does not provide audio and/or video consent, only written notes will be taken. F&P Nasal efficacy data will be downloaded from participants' PAP/BPAP therapy devices. If the participant prefers their usual mask over the F&P Nasal mask, they will return the F&P Nasal mask and the User Instruction (UI) and return to using their usual mask and will be considered to have completed the investigation.

If the participants prefer the F&P Nasal mask to their usual mask they will be invited to continue to use the F&P Nasal mask in-home for an additional 6 months. Monthly phone calls will be made and recorded in the CRF and at the end of six months the participants will be asked to return the mask and UI to CSI and provide their feedback in the form of verbal comments and a structured questionnaire (Appendix B). This will mark the 4<sup>th</sup> Visit and end of the extension part of the trial. Participants will return the F&P Nasal mask, and continue using their usual mask.

This study will be conducted in accordance with ICH/GCP Guidelines. No deviation from the protocol will be implemented without the prior review and approval of the sponsor except where it may be

necessary to eliminate an immediate hazard to a research participant. In such case, the deviation will be reported to the sponsor as soon as possible.

### 6.2. Literature Review

Obstructive Sleep Apnea (OSA) is a common sleep breathing disorder ranging from 9% to 38% in the general adult population<sup>3</sup> and is characterized by periodic collapse of the upper airway during sleep. The standard treatment for obstructive sleep apnea is PAP, which consists of pressurized air applied to the nose via an interface. PAP includes continuous positive airway pressure (CPAP), automatic positive airway pressure (APAP) and Bilevel positive airway pressure (BPAP). Despite the effectiveness of PAP in abolishing upper airway obstruction, acceptance of and adherence with therapy has been sub-optimal<sup>4,5</sup>. Reasons for the low compliance include nocturnal awakenings, incorrect therapeutic pressure and primarily discomfort due to poor mask fit. Poor mask fit can result in facial abrasion, leak causing fluctuations in therapeutic pressure and irritation of the eyes<sup>6,7</sup>.





### 6.5. Justification for Administration

Participants will remain on their prescribed PAP /BPAP therapy pressures and devices during the duration of the trial. Baseline PAP /BPAP therapy data on the participant's usual mask will be collected after  $7 \pm 3$  days in order to evaluate treatment efficacy compared to the investigational mask. Participants will not be randomised to use the F&P Nasal in-home for  $14 \pm 3$  days.

# 7. Objectives of the Clinical Investigation

### 7.1. Hypothesis

### 7.2. Objectives

Primary Objective:

 To evaluate the performance, comfort and ease of use (usability) of the F&P Nasal mask in a home environment in regards to the participants' view on overall comfort, overall experience and satisfaction.

### Secondary Objective:

 To evaluate the performance, comfort and ease of use (usability) of the F&P Nasal mask in a home environment in regards to the participants' view on overall comfort, overall experience and satisfaction over time.

### 7.3. Population

This investigation is a prospective, randomized, non-blinded study. This investigation is designed to evaluate the performance, comfort and ease of use of the F&P Nasal mask amongst a minimum of 45 participants diagnosed with OSA who are current nasal, sub-nasal or pillows users.



## 7.6. Type of Investigation

This is an open-label (investigators and participants are non-blinded and informed of intended treatment device) single arm study. The F&P Nasal will provide effective treatment similar to the



participant's usual CPAP mask. The intended treatment F&P Nasal will not be randomized – as the intention is not to compare between masks therapies.

### 7.7. Controls

The PAP/BPAP therapy device data gathered from the participants using their usual mask at baseline will act as the control for each participant, and will be compared to the data gathered from participants when using the F&P Nasal mask.

### 7.8. Bias

The F&P Nasal mask is non-blinded and distinguishable. Since the trial mask is the same for the entire population, this study is not blinded.

### 7.9. End Points

### 7.9.1. Primary Outcome

- The F&P Nasal mask provides adequate therapy for OSA during in-home use.

### 7.9.2. Secondary Outcomes

- The F&P Nasal mask is rated easy to use by the participant.
- The F&P Nasal mask is rated as comfortable to use by the participant.
- The F&P Nasal mask is rated overall by the participant as satisfactory.

### 7.10. Variables

| Variable | Justification |
|---|---|
| Ease of use/Acceptability | To assess the ease of using the mask in the home and overall mask acceptability |
| Mask Comfort | To assess the comfort (or lack of) of the mask as experienced by the participant while using it in-home. |
| Usability of the<br>mask | To evaluate the usability of the mask through a custom designed ease of use usability script |
| General<br>Demographics | To gather participants general demographics |
| Preference | To assess which mask |













### 7.12. Equipment

Participants will use their own PAP/BPAP therapy devices with their prescribed pressures.

# 7.13. Inclusion / Exclusion criteria Inclusion Criteria

- Diagnosis of OSA by Physician
- ≥ 22 years of age
- ≥ 66 lbs
- Prescribed PAP or BPAP therapy for OSA
- Existing nasal, sub-nasal and pillows mask users for approximately three months prior to enrollment in this investigation
- Fluent in written and spoken English

### **Exclusion Criteria**

- Inability to give informed consent
- Pregnant or think they may be pregnant
- PAP Intolerant
- Anatomical or Physiological Conditions that make PAP therapy inappropriate



- IPAP pressure of >25cmH20
- PAP/BPAP therapy device usage for delivery of medicines with exception of oxygen

### 7.14. Point of Enrolment

Participants will be recruited from patients who are prescribed either APAP, CPAP or BPAP devices for OSA therapy at Clayton Sleep Institute. The principal investigator (or those identified in delegation log) will ask the subjects whether they're interested to take part in the trial. The participants who provide informed consent and meet the inclusion/exclusion criteria will then be enrolled into the trial.

### 7.15. Patient Procedure

The study coordinator will ask the subjects whether they're interested to take part in the trial. Only eligible participants, that provide written informed consent, will be enrolled into the investigation.

| EVENTS | Visit<br>One | Visit<br>Two | Phone<br>Call | Visit<br>Three | Phone call | Phone call | Phone call | Phone call | Phone call | Visit<br>Four |
|---|---|---|---|---|---|---|---|---|---|---|
| Informed consent<br>(CIA-262) | X | | | | | | | | | |
| Commence baseline data gathering | Х | | | | | | | | | |
| Participant<br>Questionnaire (see<br>Appendix B) | Х | Х | | | | | | | | |
| Mask fitting with F&P Nasal mask | | Х | | | | | | | | |
| Static Leak<br>Measurement | | Х | | | | | | | | |
| Issue complete<br>Nasal<br>mask with UI | | X | | | | | | | | |
| Sleep Diary Issued | | X | | | | | | | | |
| Researcher<br>Questionnaire (see<br>Appendix C) | | X | | Х | | | | | | |
| Baseline PAP<br>device data<br>downloaded | | Х | | | | | | | | |
| Commence in-home trial of the F&P | | Х | | | | | | | | |

| EVENTS | Visit<br>One | Visit<br>Two | Phone<br>Call | Visit<br>Three | Phone call | Phone call | Phone call | Phone call | Phone call | Visit<br>Four |
|---|---|---|---|---|---|---|---|---|---|---|
| Nasal mask | | | | | | | | | | |
| Phone call | | | X | | | | | | | |
| Return the F&P<br>Nasal mask | | | | Х | | | | | | |
| PAP device data downloaded | | Х | | Х | | | | | | |
| AE/SAE assessment | | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Commence F&P<br>Nasal extension if<br>participant agrees | | | | X | | | | | | |
| Phone call (extension month 1) | | | | | Х | | | | | |
| Phone call (extension month 2) | | | | | | Х | | | | |
| Phone call (extension month 3) | | | | | | | Х | | | |
| Phone call (extension month 4) | | | | | | | | Х | | |
| Phone call (extension month 5) | | | | | | | | | Х | |
| PAP device data downloaded | | | | | | | | | | Х |
| Return F&P Nasal mask. | | | | | | | | | | Х |
| Participant<br>Questionnaire (see<br>Appendix B) | | | | | | | | | | Х |







| With the following section, the days $(\pm N)$ reflects: the date that will begin for within which the visit is acceptable) | that section (± the range |
|---|---|





### 7.16. Withdrawal Criteria

Participants will be informed that they have the right to withdraw from the study at any time, without prejudice to their medical care, and are not obliged to state their reasons. The participants are informed that they can revert back to their usual therapy during the clinical investigation if they have reason to do so. Additionally the investigator may withdraw a participant at any time for the following reasons:

- Protocol Violation
- Safety concerns
- Serious illness
- Adverse event

The reason for participant discontinuation in the study is to be recorded in the CRF and source document.

### 7.17. Number of Trial Subjects

A minimum of 45 nasal, sub-nasal and pillows mask users for OSA therapy will be recruited into this trial.

### 7.18. Follow up Plan

Participants will receive standard care from their health care provider throughout and following the study.



Since the trial is regarding the performance and acceptability of the trial device in order to inform product development, no statistical design is required.





### 7.22. Statistical Termination

No interim analysis will be conducted as statistical outcomes will not change the conduct of the study.

### 7.23. Statistical Procedure Deviations

Statistical procedure deviations will be reported to the principal investigator and the sponsor. Deviations from the original statistical plan will be explained in the final study report.

### 7.25. Statistical Data Management

Fisher and Paykel Healthcare may consult an external statistician to assist with the analysis of the data.

### 8. Adverse Events and Termination

An Adverse Event (AE) is any adverse change from the participant's baseline condition, i.e., any unfavourable and unintended sign or symptom or disease that occurs during the course of the study, whether or not considered related to the PAP treatment. All clinically significant AE's occurring during the study will be assessed at each subsequent visit and phone call to assess any change to the subject's health status since the previous interaction. Any change in health status will be recorded on CRF and evaluated by the PI.

Serious AE's are considered to be AE's that result in any of the following outcomes, regardless of their relationship to the PAP treatment:

- Death
- A life-threatening AE
- In-patient hospitalization or prolongation of existing hospitalization
- A persistent or significant disability/incapacity
- A congenital abnormality/birth defect





### 8.3. Reporting Adverse Events

Any serious AE, due to any cause, that occurs during the study period, must be reported immediately (within the next business day) by telephone to the sponsor. In addition to the initial telephone report, a Serious Adverse Event form must be completed and sent via facsimile to the sponsor. All serious AE's must also be recorded on the AE page of the CRF. Additionally, all serious AE's must be reported to the Independent Review Board (IRB) as per the IRB's requirements.



### 8.4. Early Termination

The study may be discontinued at any time on the advice of the responsible investigator on the basis of new information regarding safety or efficacy. Additionally, the study may be terminated if progress is unsatisfactory.

The following documentation is required if the appropriate party terminates a clinical trial.

### 8.4.1. Investigator

If the investigator terminates or suspends a trial without prior agreement of the sponsor, the investigator should inform the institution, where required by the applicable regulatory requirements and the investigator/institution should promptly inform the sponsor and the IRB, and should provide the sponsor and the IRB a detailed written explanation of the termination or suspension.

### 8.4.2. Sponsor

If the sponsor terminates or suspends a trial, the investigator should promptly inform the institution, where required by the applicable regulatory requirements, and the investigator/institution should promptly inform the IRB and provide the IRB a detailed written explanation of the termination or suspension.

### 8.4.3. Institutional Review Board (IRB) or Independent Ethics Committee (IEC)

If the IRB terminates or suspends its approval/favorable opinion of a trial the investigator should inform the institution, where required by the applicable regulatory requirements, and the investigator/institution should promptly notify the sponsor and provide the sponsor with a detailed written explanation of the termination or suspension.

# 9. Publication Policy

This study is intended for internal use on the development of the product. However the results of this study may be used for marketing purposes or in regulatory documentation to support the clinical efficacy of the devices.

# 10. Approval

All the required signatories for the approval of this document (Clinical Investigation Plan) are listed on the front page of this document with their relevant positions. Signing the below approval indicates that the primary investigator (PI) agrees to this version of CIP.





### 11. References

- Schein AS, Kerkhoff AC, Coronel CC, Plentz RD, Sbruzzi G. Continuous positive airway pressure reduces blood pressure in patients with obstructive sleep apnea; a systematic review and meta-analysis with 1000 patients. J Hypertens. 2014;32(9):1762–73.
- 2. Marshall NS, Barnes M, Travier N, Campbell AJ, Pierce RJ, McEvoy RD, et al. Continuous positive airway pressure reduces daytime sleepiness in mild to moderate obstructive sleep apnoea: a meta-analysis. Thorax. 2006;61(5):430–4.
- 3. Senaratna CV, Perret JL, Lodge C, Lowe A, Campbell BE, Matheson MC, Hamilton GS, Dharmage SC, Prevalence of Obstructive Sleep Apnea in the general population: A systematic review, *Sleep Medicine Reviews* (2016).
- 4. Dungan G et al. Randomized Crossover Trial of the Effect of a Novel Method of Pressure Control (SensAwake) in Automatic Continuous Positive Airway Pressure Therapy to Treat Sleep Disordered Breathing. Journal of Clinical Sleep Medicine 2011; 7(3): 261-267.
- 5. Kribbs NB et al. Objective measurement of patterns of nasal CPAP use by patients with obstructive sleep apnea. Am Rev Respir Dis 1993; 147(4): 887-95.
- 6. Weaver T, Grunstein T (2008) Adherence to continuous positive airway pressure: the challenge to effective treatment. Proc Am Thorac Soc 15(5):173–178.
- 7. Wolkove N, Baltzan M, Kamel H, Dabrusin R, Palayew M (2008) Long-term compliance with continuous positive airway pressure in patients with obstructive sleep apnea. Can Respir J 15(7):365–369.
- 8. Massie CA and Hart RW. Clinical Outcomes related to Interface type in patients with Obstructive Sleep Apnea/Hypopnea Syndrome who are using Continuous Positive Airway Pressure. Chest 2003; 123:1112-1118.
- 9. Elliott MW. The Interface: crucial for successful non-invasive ventilation. European Respiratory Journal 2004; 23:7-8.
- 10. Schnohofer B and Sortor-Leger S. Equipment needs for non-invasive mechanical ventilation. European Respiratory Journal 2002; 20:1029-1036.
- 11. Scharf S et al. Racial Differences in Clinical Presentation of patients with Sleep-Disordered Breathing. Sleep and Breathing 2004; 8(4): 173-183.
- 12. Meetze K et al. Obstructive Sleep Anea: A Comparison of Black and White Subjects. The Laryngoscope 2002; 112(7):1271–1274.
- 13. Subramanian S et al. Influence of Gender and Anthropometric Measures on Severity of Obstructive Sleep Apnea. Sleep and Breathing 2012; 16(4): 1091-1095.
- 14. Davidson T, Patel M. Waist Circumference and Sleep Disordered Breathing. The Laryngoscope 2008; 118(2): 339-347.
- 15. Schwab RJ et al. An Official American Thoracic Society Statement: Continuous Positive Airway Pressure Adherence Tracking Systems: The Optimal Monitoring Strategies and Outcome Measures in Adults. Am J Respir Crit Care Med Vol 188, Iss. 5, pp 613–620, Sep 1, 2013.
- Patil SP, Ayappa IA, Caples SM, Kimoff RJ, Patel SR, Harrod CG. Treatment of adult obstructive sleep apnea with positive airway pressure: an American Academy of Sleep Medicine clinical practice guideline. *J Clin Sleep Med*. 2019;15(2):335–343.

- 17. Guy W,. ECDEU Assessment Manual for Psychopharmacology. 1976. Rockville, MD, U.S. Department of Health, Education, and Welfare.
- Baltzan MA, Dabrusin R, Garcia-Asensi A, Sully J-L, Parenteau M, Tansimat G, et al. Leak Profile Inspection During Nasal Continuous Positive Airway Pressure. Respir Care. 2011 May;56(5):591 LP-595.
- 19. Teschler H, Stampa J, Ragette R, Konietzko N, Berthon-Jones M. Effect of mouth leak on effectiveness of nasal bilevel ventilatory assistance and sleep architecture. Eur Respir J. Eur Respiratory Soc; 1999;14(6):1251–7.
- 20. Morgenthaler TI, Aurora RN, Brown T, Zak R, Alessi C, Boehlecke B, et al. Practice parameters for the use of autotitrating continuous positive airway pressure devices for titrating pressures and treating adult patients with obstructive sleep apnea syndrome: an update for 2007. An American Academy of Sleep Medicine report. Sleep [Internet]. Associated Professional Sleep Societies, LLC; 2008 Jan 1;31(1):141–7.
- 21. Applying Human Factors and Usability Engineering to Medical Devices: Guidance for Industry and Food and Drug Administration (FDA) staff. Issued on 03 February 2016.




































































